CLINICAL TRIAL: NCT04109079
Title: ATNEC - Axillary Management in T1-3N1M0 Breast Cancer Patients With Needle Biopsy Proven Nodal Metastases at Presentation After Neoadjuvant Chemotherapy
Brief Title: Axillary Management in Breast Cancer Patients With Needle Biopsy Proven Nodal Metastases After Neoadjuvant Chemotherapy
Acronym: ATNEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Amit Goyal, Consultant Oncoplastic Breast Surgeon & Associate Professor, University Hospitals of Derby and Burton NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIHR 128311
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Sentinel Lymph Node; Neoplasm, Breast
Keywords: neoadjuvant chemotherapy; sentinel node biopsy; breast cancer; tattooing node; marking node; clip node; axillary ultrasound; node positive; axillary lymph node dissection; axillary radiotherapy; axillary treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No axillary treatment (Experimental): Patients in this arm will not receive axillary treatment (axillary lymph node dissection or axillary radiotherapy). Supraclavicular fossa radiotherapy is not allowed when randomised to this arm.
  Interventions: Radiation: Breast or chest wall radiotherapy
- Axillary treatment (Active Comparator): Patients in this arm will receive axillary treatment. Axillary treatment can be axillary lymph node dissection or axillary radiotherapy.
  Interventions: Procedure: Axillary lymph node dissection; Radiation: Axillary radiotherapy; Radiation: Breast or chest wall radiotherapy

INTERVENTIONS:
Procedure: Axillary lymph node dissection — Participants will undergo removal of at least level I and II axillary lymph nodes.
  Arms: Axillary treatment
Radiation: Axillary radiotherapy — Axillary radiotherapy will be delivered as per the Radiotherapy Trials Quality Assurance (RTTQA) guidelines.
  Arms: Axillary treatment
Radiation: Breast or chest wall radiotherapy — Breast or chest wall radiotherapy will be delivered as per the Radiotherapy Trials Quality Assurance (RTTQA) guidelines.

SUMMARY:
The aim of this study is to assess whether, omitting further axillary treatment (ALND and ART) for patients with early stage breast cancer and axillary nodal metastases on needle biopsy, who after NACT have no residual cancer in the lymph nodes on sentinel node biopsy, is non-inferior to axillary treatment in terms of disease free survival (DFS) and results in reduced risk of lymphoedema at 5 years.

DETAILED DESCRIPTION:
Background: The presence of cancer in the axillary lymph nodes on needle biopsy in patients with early stage breast cancer before neoadjuvant chemotherapy (NACT) has been the determinant of the need for axillary treatment (in the form of axillary lymph node dissection (ALND) or axillary radiotherapy (ART)) after completion of NACT. Treatment to the axilla damages lymphatic drainage from the arm and patients can subsequently develop lymphoedema, restricted shoulder movement, pain, numbness, and other sensory problems. As more effective chemotherapy is now available that results in complete eradication of cancer in the axilla in around 40 to 70% of patients, extensive axillary treatment might no longer be necessary in patients with no evidence of residual nodal disease.

Aim: To assess whether, omitting further axillary treatment (ALND and ART) for patients with early stage breast cancer and axillary nodal metastases on needle biopsy, who after NACT have no residual cancer in the lymph nodes on sentinel node biopsy, is non-inferior to axillary treatment in terms of disease free survival (DFS) and results in reduced risk of lymphoedema at 5 years.

Methods:

Study design: A pragmatic, phase 3, open, randomised, multicentre trial and embedded economic evaluation in which participants will be randomised in a 1:1 ratio.

Study population: T1-3N1M0 breast cancer patients aged 18 years or older, with needle biopsy proven nodal metastases, who after NACT have no residual cancer in the lymph nodes on dual tracer sentinel node biopsy and removal of at least 3 lymph nodes (sentinel nodes and marked involved node).

Intervention: All participants will receive human epidermal growth factor receptor 2 (HER2)-targeted treatment, endocrine therapy and radiotherapy to breast or chest wall, if indicated according to local guidelines. Patients in the intervention group will not receive further axillary treatment (ALND or ART), whereas those receiving standard care will receive axillary treatment (ALND or ART) as per local guidelines. Follow-up is annually for at least 5 years.

Outcomes: The co-primary outcomes are disease free survival(DFS) and self-reported lymphoedema defined as 'yes' to the two questions participants will be asked - 'arm heaviness during the past year' and 'arm swelling now' from the Lymphoedema and Breast Cancer Questionnaire at 5 years.

Secondary outcomes: arm function assessed by the QuickDASH (disabilities of the arm, shoulder and hand) questionnaire; health related quality of life assessed using euroqol EQ-5D-5L; axillary recurrence free interval (ARFI); local recurrence; regional (nodal) recurrence; distant metastasis; overall survival; contralateral breast cancer; non-breast malignancy; costs; quality adjusted life years (QALYs) and cost-effectiveness.

Sample size: A sample size of 1900 patients would have the ability to demonstrate a 3.5% non-inferiority margin with a 5% 1-sided significance level and 85% power, allowing for 7% non-collection of primary outcome data assuming a 90% 5-year disease free survival rate in the control arm. It would also be able to detect at least a 5% difference in proportion of patients with lymphoedema with 90% power, a 5% 2-sided significance level and allowing for 25% non-collection of primary outcome data over 5 years.

Analysis plan: All analyses will be carried out on an intention-to-treat basis to preserve randomisation, avoid bias from exclusions and preserve statistical power. Time to event outcomes, including disease free survival and axillary recurrence free interval, will be assessed using Kaplan-Meier curves and compared using Cox proportional hazards models. The proportion of patients experiencing lymphoedema at 5 years will be compared across trial arms using a chi-squared test and a logistic regression model used to adjust for stratification variables. Arm morbidity and health related quality of life will be scored using the appropriate manuals and assessed using a longitudinal mixed model regression analysis if model assumptions valid or a standardised area-under-the-curve analysis. For economic evaluation, incremental cost per QALY gained at 5 years will be estimated.

Timelines for delivery: Total project duration is 120 months based on 6 months for set up; 60 months recruitment period (including an 18 months internal pilot phase); and 54 months for follow up, analysis, writing up and dissemination.

ELIGIBILITY:
Inclusion Criteria:

* cT1-3N1M0 breast cancer at diagnosis (prior to NACT) by American Joint Committee on Cancer (AJCC) staging 8th edition
* Patients with occult primary breast cancer (no identifiable invasive cancer in the breast) with FNA or core biopsy proven nodal metastases are also eligible for the study.
* Fine-needle aspiration (FNA) or core biopsy confirmed axillary nodal metastases at presentation
* Oestrogen receptor and HER2 status evaluated on primary tumour
* Received standard NACT as per local guidelines (Patients undergoing neoadjuvant endocrine therapy as part of another clinical trial are eligible)
* Imaging of the axilla, as required, to assess response to NACT (per local guidelines)
* Undergo a dual tracer sentinel node biopsy (SNB) after NACT with at least 3 nodes removed in total (sentinel nodes and marked node).
* If a single tracer SNB is performed, the patient is eligible only if the involved node is marked before or during NACT, and at least 3 nodes (including the marked node) are removed during sentinel node biopsy.
* If the node is not marked, or the marked node is not removed, the patient is eligible only if the histology report shows evidence of down-staging with complete pathological response e.g. fibrosis or scarring in at least one node and at least 3 nodes removed.
* If fewer than 3 nodes are found on histology, the patient is eligible only if BOTH points a) and b) below, are met:

  1. involved node was marked and removed during SNB; and
  2. removed marked node shows evidence of downstaging on histology e.g. fibrosis or scarring.
* If the sentinel node(s) cannot be localised on SNB: axillary node sampling should be performed, the patient will be eligible if at least 3 nodes are removed (including the marked node).
* No evidence of nodal metastases post NACT (isolated tumour cells, micro or macro metastasis)
* Patients with complete pathological response in the axilla but residual disease in the breast post NACT are eligible for the study.

Exclusion Criteria:

* Bilateral synchronous invasive breast cancer
* Sentinel node biopsy prior to NACT
* Previous axillary surgery on the same body side as the scheduled targeted sampling
* Any previous cancer within 5 years or concomitant malignancy except

  * basal or squamous cell carcinoma of the skin
  * in situ carcinoma of the cervix
  * in situ melanoma
  * contra- or ipsilateral in situ breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) | 5 years
  DFS calculated as the time from randomisation until the date of first event of either a loco-regional invasive breast cancer relapse, distant relapse, ipsilateral or contralateral new invasive primary breast cancer or death by any cause or the censor date.
Patient reported lymphoedema | 5 years
  Lymphoedema is self-reported based on two items from the validated Lymphoedema and Breast Cancer Questionnaire (arm "swelling now" and arm "heaviness in the past year"). Lymphoedema is defined as 'yes' to both questions.

SECONDARY OUTCOMES:
Arm function | 5 years
  Arm function will be assessed using shortened version of the Disability of the Arm, Shoulder and Hand (DASH), the 11-item QuickDASH questionnaire. Physical disability is defined as a change from baseline in the QuickDASH score of at least 14 points.
Health related quality of life: EQ-5D-5L | 5 years
  Health related quality of life will be assessed with EQ-5D-5L
Axillary recurrence free interval | 5 years
  Axillary recurrence free interval, calculated from the date of randomisation to the date of axillary recurrence or the censor date.
Overall survival | 5 years
  Overall survival calculated as the time from randomisation until the date of death by any cause or the censor date.
Local (breast or chest wall) recurrence | 5 years
  Number of participants with local (breast or chest wall) recurrence
Regional (nodal) recurrence | 5 years
  Number of participants with regional (nodal) recurrence
Distant metastasis | 5 years
  Number of participants with distant metastasis.
Contralateral breast cancer | 5 years
  Number of participants with contralateral breast cancer.
Non-breast cancer | 5 years
  Number of participants with non-breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Amit Goyal, MS, MD, FRCS, Principal Investigator — Royal Derby Hospital, Derby, UK
Locations (98):
- Ireland (4):
  - St Vincent's University Hospital - St Vincent's Healthcare Group, Dublin
  - St Luke's Hospital - St Luke's Radiation Oncology Network, Dublin
  - Beaumont Hospital - Royal College of Surgeons in Ireland, Dublin
  - Galway University Hospitals - Saolta University Health Care Group, Galway
- United Kingdom (94):
  - Airedale General Hospital - Airedale NHS Foundation Trust, Keighley, BD20 6TD
  - Cumberland Infirmary - North Cumbria Integrated Care NHS Foundation Trust, Carlisle, CA2 7HY
  - Frimley Park Hospital - Frimley Health NHS Foundation Trust, Camberley, GU16 7UJ
  - Raigmore Hospital - NHS Highland, Inverness, IV2 3UJ
  - James Paget Hospital -James Paget University Hospitals NHS Foundation Trust, Great Yarmouth, NR31 6LA
  - Royal Berkshire Hospital - Royal Berkshire NHS Foundation Trust, Reading, RG1 5AN
  - Macclesfield District General Hospital - East Cheshire NHS Trust, Macclesfield, SK10 3BL.
  - Royal Shrewsbury Hospital -The Shrewsbury and Telford Hospitals NHS Trust, Shrewsbury, SY3 8XQ
  - Aberdeen Royal Infirmary - NHS Grampian, Aberdeen
  - Ashford Hospital - Ashford and St Peter's Hospitals NHS Foundation Trust, Ashford
  - Tameside General Hospital- Tameside and Glossop Integrated Care NHS Foundation Trust, Ashton-under-Lyne
  - University Hospital Crosshouse - NHS Ayrshire and Arran, Ayr
  - Basildon University Hospital - Mid and South Essex NHS Foundation Trust, Basildon
  - Belfast City Hospital - Belfast Health and Social Care Trust, Belfast
  - QEHB- University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - City Hospital -Sandwell and West Birmingham NHS Trust, Birmingham
  - Blackpool Victoria Hospital - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - Royal Bolton Hospital - Bolton NHS Foundation Trust, Bolton
  - St Luke's Hospital - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - Royal Sussex County Hospital - University Hospitals Sussex NHS Foundation Trust, Brighton
  - Southmead Hospital - North Bristol NHS Trust, Bristol
  - Burnley General Hospital- East Lancashire Hospitals NHS Trust, Burnley
  - Addenbrooke's Hospital - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cheltenham General Hospital - Gloucestershire General Hospitals NHS Foundation Trust, Cheltenham
  - Countess of Chester Hospital - Countess of Chester Hospital NHS Trust, Chester
  - Leighton Hospital - Mid Cheshire NHS Foundation Trust, Crewe
  - Darlington Memorial Hospital - County Durham and Darlington NHS Foundation Trust, Darlington
  - Royal Derby Hospital- University Hospitals of Derby and Burton NHS Foundation Trust, Derby
  - Doncaster Royal Infirmary - Doncaster and Bassetlaw Teaching Hospitals NHS Foundation Trust, Doncaster
  - Russell's Hall Hospital - The Dudley Group NHS Foundation Trust, Dudley
  - Dumfries and Galloway Royal Infirmary - NHS Dumfries and Galloway, Dumfries
  - Queen Margert Hospital - NHS Fife, Dunfermline
  - University Hospital Hairmyres - NHS Lanarkshire, East Kilbride
  - Western General Hospital -NHS Lothian, Edinburgh
  - Royal Devon & Exeter Hospital - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Queen Elizabeth Hospital - Gateshead Health NHS Foundation Trust, Gateshead
  - Beatson West of Scotland Cancer Centre - Greater Glasgow Health Board, Glasgow
  - Royal Surrey County Hospital - Royal Surrey NHS Foundation Trust, Guildford
  - Harrogate District Hospital - Harrogate and District NHS Foundation Trust, Harrogate
  - Hereford County Hospital- Wye Valley NHS Trust, Hereford
  - Wycombe Hospital - Buckinghamshire Healthcare NHS Trust, High Wycombe
  - Huddersfield Royal Infirmary- Calderdale and Huddersfield NHS Foundation Trust, Huddersfield
  - Castle Hill Hospital - Hull University Teaching Hospitals NHS Trust, Hull
  - Ipswich Hospital - East Suffolk and North Essex NHS Foundation Trust, Ipswich
  - West Middlesex University Hospital - Chelsea and Westminster Hospital NHS Foundation Trust, Isleworth
  - Royal Lancaster Infirmary - University Hospitals of Morecambe Bay NHS Foundation Trust, Lancaster
  - Forth Valley Royal Hospital - NHS Forth Valley, Larbert
  - St James's University Hospital - Leeds Teaching Hospitals NHS Trust, Leeds
  - Glenfield Hospital - University Hospitals of Leicester NHS Trust, Leicester
  - Lincoln County Hospital - United Lincolnshire Hospitals NHS Trust, Lincoln
  - Prince Phillip Hospital -Hywel Dda University Health Board, Llanelli
  - North Middlesex University Hospital - North Middlesex University Hospital NHS Trust, London
  - The Whittington Hospital - Whittington Health NHS Trust, London
  - UCL Hospital - University College London Hospitals NHS Foundation Trust, London
  - Royal Free Hospital - Royal Free London NHS Foundation Trust, London
  - Kings College Hospital - King's College Hospital NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - Charing Cross Hospital -Imperial College Healthcare NHS Trust, London
  - Luton and Dunstable Hospital -Bedfordshire Hospitals NHS Foundation Trust, Luton
  - Wythenshawe Hospital - Manchester University Hospital NHS Foundation Trust, Manchester
  - North Manchester General -Manchester University NHS Foundation Trust, Manchester
  - Borders General Hospital -NHS Borders, Melrose
  - Clatterbridge Cancer Centre - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Clatterbridge Hospital - Wirral University Teaching Hospital NHS Foundation Trust, Metropolitan Borough of Wirral
  - The James Cook University Hospital - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Milton Keynes Hospital - Milton Keynes University Hospital NHS Trust, Milton Keynes
  - Royal Victoria Infirmary- Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - North Tyneside General Hospital - Northumbria Healthcare NHS Foundation Trust, North Shields
  - Churchill Hospital - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Royal Alexandra Hospital - NHS Greater Glasgow and Clyde, Paisley
  - Derriford Hospital - University Hospitals Plymouth NHS Trust, Plymouth
  - Queen Alexandra Hospital - Portsmouth Hospitals University NHS Trust, Portsmouth
  - St Helen's Hospital - St Helens and Knowsley Teaching Hospitals NHS Trust, Prescot
  - Royal Preston Hospital - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - East Surrey Hospital - Surrey & Sussex Healthcare NHS Trust, Redhill
  - Rotherham General Hospital - The Rotherham NHS Foundation Trust, Rotherham
  - Weston Park Hospital - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - St Alban's Hospital - West Hertfordshire Hospitals NHS Trust, St Albans
  - Lister Hospital - East and North Hertfordshire NHS Foundation Trust, Stevenage
  - University Hospital North Tees - North Tees and Hartlepool NHS Foundation Trust, Stockton-on-Tees
  - Royal Stoke University Hospital - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent
  - Singleton hospital - Swansea Bay University Health Board, Swansea
  - Musgrove park Hospital -Somerset NHS Foundation Trust, Taunton
  - Croydon University Hospital - Croydon Health Services NHS Trust, Thornton Heath
  - Royal Cornwall Hospital - Royal Cornwall Hospitals NHS Trust, Truro
  - Hillingdon Hospital - The Hillingdon Hospitals NHS Foundation Trust, Uxbridge
  - Pinderfields Hospital - Mid Yorkshire Hospitals NHS Trust, Wakefield
  - Southend Hospital and Broomfield Hospital -Mid and South Essex NHS Foundation Trust, Westcliff-on-Sea
  - Royal Albert Edward Infirmary - Wrightington, Wigan and Leigh Teaching Hospitals NHS Foundation Trust, Wigan
  - King Edward VII Hospital - Frimley Health NHS Foundation Trust, Windsor
  - New Cross Hospital - The Royal Wolverhampton NHS Trust, Wolverhampton
  - Worcestershire Royal Hospital - Worcestershire Acute Hospitals NHS Trust, Worcester
  - Yeovil District Hospital -Yeovil District Hospital NHS Trust, Yeovil
  - York Hospital - York and Scarborough Teaching Hospitals NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Training video for surgeons to remove the marked node during sentinel node biopsy — https://youtu.be/SFAzvkpkM84
- See also: Training video for radiologists to mark the node using black dye tattoo — https://youtu.be/Nq3tmI6l66s
- See also: Training video for radiologists to mark the node using clip — https://youtu.be/nLA0fYihVOc
- See also: ATNEC breast cancer study - Research Nurse and Patient Consultation — https://www.youtube.com/watch?v=s5vqST08HYE
- See also: ATNEC breast cancer study - Example Doctor and Patient Consultation — https://www.youtube.com/watch?v=0zAl4PkJV-w&t=4s